CLINICAL TRIAL: NCT03813693
Title: Surgical Site Infection and the Use of 2% Chlorhexidine Gluconate Impregnated Cloth Bathing in Preoperative Skin Preparation: a Pilot Randomized Clinical Trial.
Brief Title: The Use of 2% Chlorhexidine Gluconate Impregnated Cloth Bathing in Preoperative Skin Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernanda de Oliveira Andrade, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EEUSP
Record Dates: First submitted 2019-01-09; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: The intervention group (GI) received two packs, each containing six towels impregnated with 2% chlorhexidine gluconate and an instruction manual on how to use them.
  Two bottles of chlorhexidine gluconate 2% liquid (100 ml) were given to the control group (CG), the patients were instructed to perform the bath using one vial the night before surgery and the other on the morning of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- towels with chlorhexidine gluconate 2% (Experimental): Composed of 25 patients, who received 2 towels with chlorhexidine gluconate 2% packages each containing six towels and detailed instructions on the form and sequence of application of the towels; the time of application, that is, the night before surgery, between 20 and 22h, and, on the morning of surgery, between 5 and 6h; besides other general orientations.
  Interventions: Other: towels impregnated with 2% chlorhexidine gluconate
- chlorhexidine gluconate 2% liquid (Active Comparator): Composed of 23 patients, two 100 ml flasks of chlorhexidine gluconate 2% liquid were supplied, and detailed instruction manual for the product, containing form and application sequence; time of application (the night before surgery, between 20 and 22h, and on the morning of surgery, between 5 and 6h); and general guidelines.
  Interventions: Other: chlorhexidine gluconate 2% liquid

INTERVENTIONS:
Other: towels impregnated with 2% chlorhexidine gluconate — The first TICHG should be used on the neck, chest and abdomen; The second TICHG should be used on the right upper limb, start at the shoulder; The third TICHG was intended for the upper left limb; The fourth TICHG should be used on the neck and chest; The fifth TICHG was for the right lower limb; The sixth TICHG should be used on the lower left limb.
  2) Time of application: use six TICHGs the night before surgery and the six remaining on the morning of surgery.
  3) After the hygiene of each member, discard the TICHG. After use of TICHG, allow the product to dry on the skin. Do not use bath towels to dry yourself and wear clean clothes.
  Arms: towels with chlorhexidine gluconate 2%
Other: chlorhexidine gluconate 2% liquid — Spread the product on the skin during the bath and massage for 3 minutes, so that it is distributed equally to all parts of the body (except the face, hair and intimate area). Then rinse with water and dry with a clean, dry towel, and wear clean clothes.
  Arms: chlorhexidine gluconate 2% liquid

SUMMARY:
To compare the use of towels impregnated with 2% chlorhexidine gluconate in the traditional preoperative bath with 2% chlorhexidine gluconate in preventing the occurrence of surgical site infection among patients undergoing potentially contaminated elective surgery.

DETAILED DESCRIPTION:
This is a pilot randomized controlled clinical trial, composed of patients submitted to potentially contaminated elective surgeries, randomly assigned to an intervention group, consisting of those who used towels impregnated with pre-operative CHG 2% and control group, composed of by the pre-operative bath with 2% conventional / liquid CHG. Both used the products the night before and the morning of surgery and received verbal and written guidance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* literate
* undergoing potentially contaminated elective surgeries
* admitted on the day before the surgical treatment or in the triple three-day hospital stay prior to surgery, without an infectious or otherwise infected process
* correctly follow the instructions for the use of towels impregnated with chlorhexidine gluconate 2%
* follow the instructions for the use of chlorhexidine gluconate 2%

Exclusion Criteria:

* submitted to previous surgeries, in a period of less than thirty days, or ninety days in the case of a prosthesis implant
* present skin lesions or known allergy to chlorhexidine gluconate 2%
* patients submitted to videolaparoscopic surgeries and vaginal surgeries
* patients who had daily use of products containing antiseptics (creams and / or liquid or bar soaps containing CHG, triclosan or similar) in their daily activity; or who had used antibiotics or similar drugs two weeks before and during the period of data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Prevention of surgical site infection - Criteria: Centers for Disease Control and Prevention, 2018 | 1 month (30 days)
  In order to investigate the potential cases of SSI, the researcher personally followed the patients in the preoperative period, in the POI and at the time of hospital discharge, using a data collection instrument. In order to evaluate the occurrence of SSI after hospital discharge, the researcher used the following strategies: a review of the chart associated with patient follow-up during outpatient return when possible, which would occur on average on the 35th postoperative day; telephone contact from the 30th day until the 40th postoperative day (PO), using a post-discharge surveillance instrument. Continuous and discrete quantitative variables were evaluated using the Wilcoxon-Mann-Whitney test.
  Qualitative (categorical) variables were evaluated using the Pearson X² test. The Wilcoxon-Mann-Whitney test was used for qualitative (categorical) variables, whose distribution was different from normal.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Andrade, Principal Investigator — University of Sao Paulo; Vanessa Poveda, Principal Investigator — University of Sao Paulo
Locations (1):
- Fernanda de Oliveira Andrade, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No